CLINICAL TRIAL: NCT04209647
Title: A Comparison of Reduced HIIT and Moderate Intensity Continuous Exercise in Obese Young Adults
Brief Title: A Comparison of Continuous Moderate Training and Reduced High Intensity Interval Training in Obese Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Associate Proffesor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0004
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Exercise; Oxygen Consumption
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Exercise (Active Comparator): At %60 of maximal heart rate, 30-60 minutes exercise
  Interventions: Other: Continuous Aerobic Exercise
- REHIT Exercise (Experimental): At %100 of heart rate 15 seconds, after this period 15 sec recovery period for all step
  Interventions: Other: REHIT Exercise

INTERVENTIONS:
Other: REHIT Exercise — -Start with warm-up period --> %50 of maximum work rate, 3 minutes
  One Exercise Cycle consists of:
  * 15 seconds exercise period: %100 of maximum work rate
  * 15 seconds recovery period: %50 of maximum work rate
  Total Duration: 10 minutes
  Arms: REHIT Exercise
Other: Continuous Aerobic Exercise — At %50 of maximum heart rate, 30-60 minutes aerobic exercise
  Arms: Continuous Exercise

SUMMARY:
Exercise is a key component of obesity management. Obese subjects cannot attend or sustain exercise program because of increased general fatigue, dyspnea and muscle fatigue. And they feel more exertion when comparing with normal weight subjects. Reduced-exertion high-intensity interval training (REHIT) is a alternative method to continuous exercise programs. The investigators aimed comparing metabolic effects of REHIT and continuous exercise in young adults, in this study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-22,
* BMI ≥ 30,
* Female gender,

Exclusion Criteria:

* Smoking history,
* Having any metabolic disease except obesity,

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity | 1 year
  Maximum Oxygen Uptake

SECONDARY OUTCOMES:
Total Exercise Duration | 1 year
  Exercise Test Duration

OTHER OUTCOMES:
Body Fat Percentage | 1 year
  Total Body Fat Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nurgul Durustkan Elbasi, PhD, Study Chair — Istinye University; Yunus Emre Tutuneken, PT, Study Chair — Istinye University; Yasemin Cirak, Ass Prof, Principal Investigator — Istınye U; Duygu Korkem, PhD, Study Chair — University of Health science; Beyza Karaduz, MsC, Study Chair — Hacettepe University; Ebru Calik Kutukcu, PhD, Study Chair — Hacettepe University
Locations (1):
- Istınye University, Istanbul, Turkey (Türkiye)